CLINICAL TRIAL: NCT02810405
Title: Collection of Tissue Blocks or Slides From Patients With Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110190; 11-C-0190
Record Dates: First submitted 2016-06-22; First posted 2016-06-23 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Tumor; Carcinogens; Neoplasm, Benign; Benign Neoplasms; Cancer
Keywords: Sample; Storage; Molecular Profiling; Biopsy; Repository; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Patient Samples: Patients treated at NCI with available tissue samples.

SUMMARY:
BACKGROUND:

Cancer of any type is a serious disease and despite all the progress made from past research, there is still much that is poorly understood at the molecular level. Recent advances in biomedical technology platforms have emerged as critical tools for accelerating personalized medicine. The collection of human tissue specimens has been an invaluable resource for conducting translational cancer research using these developing technologies. The ultimate goal is to understand the molecular indicators of cancer development and progression. While it is ideal to be able to study clinical samples, specifically tissue biopsies, they are however precious and are often difficult to obtain in sufficient quantities or numbers to conduct proteomic or molecular profiling studies. There exists, however, a vast archive of pathologically characterized clinical samples in the form of formalin-fixed paraffin-embedded tissue blocks. The preservation of these tissue blocks and/or slides for long-term (years) storage is an important asset that aids in translational and clinical research. This protocol will describe the procedures for receiving, labeling and storing paraffin-embedded tissue blocks and/or slides until they are needed for future analysis. When blocks are ready for analysis, the requestor will then follow the IRB protocol specific to that study.

OBJECTIVE:

- To obtain tissue blocks and slides from outside pathology departments for cancer patients being treated at the Medical Oncology Branch (MOB) and Affiliates Center for Cancer Research (CCR), National Cancer Institute (NCI) in order to store them for future studies and analysis (e.g., using molecular technology platforms).

ELIGIBILITY:

- Patients suspected of having, or with biopsy proof of malignant disease will be evaluated in the Medical Oncology Branch and Affiliates Clinics, NCI.

DESIGN:

* Tissue blocks and slides will be acquired from outside pathology departments and received by the Clinical Pharmacology Program of the MOB/CCR/NCI for coding.
* Bar-coded tissue blocks and slides will then be transferred to the Laboratory of Pathology/CCR/NCI for proper long-term storage.

DETAILED DESCRIPTION:
Background

* Cancer of any type is a serious disease and despite all the progress made from past research, there is still much that is poorly understood at the molecular level.
* Recent advances in biomedical technology platforms have emerged as critical tools for accelerating personalized medicine.
* The collection of human tissue specimens has been an invaluable resource for conducting translational cancer research using these developing technologies.
* The ultimate goal is to understand the molecular indicators of cancer development and progression.
* While it is ideal to be able to study clinical samples, specifically tissue biopsies, they are however precious and are often difficult to obtain in sufficient quantities or numbers to conduct proteomic or molecular profiling studies.
* There exists, however, a vast archive of pathologically characterized clinical samples in the form of formalin-fixed paraffin-embedded tissue blocks.
* The preservation of these tissue blocks and/or slides for long-term (years) storage is an important asset that aids in translational and clinical research.
* This protocol will describe the procedures for receiving, labeling and storing paraffinembedded tissue blocks and/or slides until they are needed for future analysis.
* When blocks are ready for analysis, the requestor will then follow the IRB protocol specific to that study.

Objective

-To obtain tissue blocks and slides from outside pathology departments for cancer patients being treated at the Genitourinary Malignancies Branch (GMB) and Affiliates Center for Cancer Research (CCR), National Cancer Institute (NCI) in order to store them for future studies and analysis (e.g., using molecular technology platforms).

Eligibility

-Patients suspected of having, or with biopsy proof of malignant disease will be evaluated in the Genitourinary Malignancies Branch (GMB) and Affiliates Clinics, NCI.

Design

* This protocol is not a research study.
* Tissue blocks and slides will be acquired from outside pathology departments and received by the Clinical Pharmacology Program of the OCD/CCR/NCI for coding.
* Bar-coded tissue blocks and slides will then be transferred to the Laboratory of Pathology/CCR/NCI for proper long-term storage.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any cancer patient who is being evaluated at the National Cancer Institute with available tissue samples (blocks or slides) is eligible
* Must be able and willing to sign an informed consent for this study
* Age: greater than or equal to 18 years of age

EXCLUSION CRITERIA:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any cancer patient who is being evaluated at the NCI with available tissue samples
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
To obtain tissue blocks and slides in order to store them for future studies and analysis (e.g., using molecular technology platforms). | duration of protocol
  To obtain tissue blocks and slides from outside pathology departments for cancer patients being treated at the Genitourinary Malignancies Branch (GMB)Medical Oncology Branch (MOB) and Affiliates Center for Cancer Research (CCR), National Cancer Institute (NCI) in order to store them for future studies and analysis (e.g., using molecular technology platforms).

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Voduc D, Kenney C, Nielsen TO. Tissue microarrays in clinical oncology. Semin Radiat Oncol. 2008 Apr;18(2):89-97. doi: 10.1016/j.semradonc.2007.10.006. PMID 18314063
- [Background] Sauter G, Simon R, Hillan K. Tissue microarrays in drug discovery. Nat Rev Drug Discov. 2003 Dec;2(12):962-72. doi: 10.1038/nrd1254. No abstract available. PMID 14654795
- [Background] Blonder J, Veenstra TD. Clinical proteomic applications of formalin-fixed paraffin-embedded tissues. Clin Lab Med. 2009 Mar;29(1):101-13. doi: 10.1016/j.cll.2009.01.006. PMID 19389554
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0190.html